CLINICAL TRIAL: NCT04979234
Title: Efficacy of an Endoluminal-suturing Device (Endomina) on Severe Obstructive Sleep Apnea Syndrome : EndoSAS
Brief Title: A Single Centre, Prospective Feasibility Study to Evaluate the Efficacy of an Endoluminal-suturing Device (Endomina) on Severe Obstructive Sleep Apnea Syndrome
Acronym: EndoSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Endo Tools Therapeutics S.A. (Industry)
Responsible Party: Principal Investigator, Michael Fernandez Y Viesca, Gastroenterologist (Dr M. Fernandez), Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2020/382
Record Dates: First submitted 2021-04-13; First posted 2021-07-28 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Sleep Apnea Syndromes; Overweight and Obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Endoscopic gastric reduction
  Interventions: Device: Endomina- Endoscopic Sleeve Gastroplasty; Behavioral: Diet

INTERVENTIONS:
Device: Endomina- Endoscopic Sleeve Gastroplasty — Endoscopic gastric reduction
Behavioral: Diet — Multidisciplinary follow up

SUMMARY:
This study aims to evaluate the efficacy of an endoluminal gastric plication using an endoluminal-suturing device to improve severe OSAS in patients with a BMI above or equal to 28 kg/m² until 34.9kg/m².

DETAILED DESCRIPTION:
Obesity is one of the most critical public health burdens worldwide. Its prevalence is increasing, as well as its comorbidities. The main comorbidity of obesity on the respiratory system is the obstructive sleep apnea syndrome (OSAS). The prevalence of OSAS in the obese population is around 45%. OSAS increased cardiovascular risk and decreased quality of life. The most alterable risk factor of OSAS is obesity. Therefore, weight loss is the cornerstone of the treatment. There is some evidence of the efficacy of weight loss surgery (lap band, sleeve gastrectomy, biliary pancreatic deviation, duodenal switch, and Roux-and-Y-gastric bypass) to improve OSAS. Current recommendations suggest bariatric surgery management for patients with a BMI > 35kg/m2 and OSAS. However, most studies have limited scientific value (retrospective observational trials), and the follow-up of patients is limited, mainly due to patients' inadequate compliance. Moreover, until now, there is no reliable predictor for the percentage of reduction of AHI caused by weight loss. On the other hand, there is no approved treatment in patients presenting a BMI between 28 kg/m² to 34.9kg/m² and OSAS.

Endoscopic endoluminal approaches to address obesity have become an important topic of interest over the past decade. Endomina® (Endo Tools Therapeutics, Gosselies, Belgium) is a novel restrictive endoluminal approach. This new procedure permitted a weight loss of 29 % on average sustained at one year. This technique was not yet evaluated in patients with 28 kg/m2 ≤ BMI ≤ 34.9/m2 to improve OSAS.

The current feasibility study aims to evaluate the efficacy of an endoluminal gastric plication using an endoluminal-suturing device to improve severe OSAS in patients with above or equal to 28 kg/m², BMI until 34.9kg/m².

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* BMI between 28 to 34.9 kg/m²
* AHI ≥ 30 events/hour
* De novo CPAP user, installed within 2 months prior enrollment
* Must be able to comply with all study requirements for the duration of the study, as outlined in the protocol. This includes complying with the visit schedule as well as study-specific procedures such as clinical assessment, endoscopy, radiography, as well as laboratory investigations
* Must be able to understand and be willing to provide written informed consent;
* Had followed the multidisciplinary bariatric workup (blood analyses, dietician, psychologist and doctor appointments)

Exclusion Criteria:

* Presence of an obesity-hypoventilation syndrome defined as a PaCO2 ≥ 45 mmHg without any other respiratory disease.
* CPAP treatment failure defined as central sleep apnea occurrence under CPAP treatment or a residual AHI > 5 under optimal CPAP treatment.
* Incompliance to cPAP treatment defined as an observance to cPAP of at least 4 hours per night in average.
* Achalasia and any other esophageal motility disorders
* Current severe esophagitis (grade C and D based on Los Angeles Classification)
* Current Gastro-duodenal ulcer
* Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity;
* Hypertension: uncontrolled hypertension during the last 3 months;
* Diabetes: uncontrolled diabetes (on insulin therapy or oral therapy with Hba1c > 10%);
* TBWL >5% over the last 6 months
* Current severe renal, hepatic, pulmonary disease or cancer;
* Current gastrointestinal stenosis or obstruction
* Pregnancy, breastfeeding or willing to become pregnant in the coming 18 months
* Bariatric surgery, balloon or other endoscopic obesity-related therapy within 6 months of enrollment in this study
* Anticoagulant therapy
* Impending gastric surgery 60 days post-intervention
* Psychiatric disorder refuted after psychological evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness on OSAS | 6 months of follow up
  Proportion of patients with an apnea-hypopnea index (AHI) reduction of 50% , after the endoscopic procedure.

SECONDARY OUTCOMES:
Effectiveness on weight loss | 6 months of follow up
  Information on efficacy will be obtained by measurements of total weight loss and excess weight loss
Change of the Epworth sleepiness scale | 6 months of follow up
  Reduction of the Epworth sleepiness scale
Change of respiratory parameters | 6 months of follow up
  Increasing of FEV1 (L) (Mandatory expiratory volume in 1 second)
Change of respiratory parameters | 6 months of follow up
  Increasing of TLC (L) (Total lung capacity)
Change of respiratory parameters | 6 months of follow up
  Increasing of KCO (%) (CO diffusion)
Incidence of all adverse event | During procedure and during the 6 months of follow up
  characterized by the incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or device that are experienced by study participants

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No